CLINICAL TRIAL: NCT02280473
Title: A Safety and Efficacy Study of Refresh Optive® Gel Drops in Patients With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11193X-001
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Refresh Optive® Gel Drops (Experimental): Refresh Optive® Gel Drops; 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Interventions: Drug: Refresh Optive® Gel Drops
- REFRESH LIQUIGEL® (Active Comparator): REFRESH LIQUIGEL®; 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Interventions: Drug: REFRESH LIQUIGEL®

INTERVENTIONS:
Drug: Refresh Optive® Gel Drops — Refresh Optive® Gel Drops; 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Arms: Refresh Optive® Gel Drops
Drug: REFRESH LIQUIGEL® — REFRESH LIQUIGEL®; 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Arms: REFRESH LIQUIGEL®

SUMMARY:
This study will evaluate the safety and efficacy o fRefresh Optive® Gel Drops in patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Current use of an artificial tear product
* Visual acuity of at least 20/32 (while wearing glasses, if necessary).

Exclusion Criteria:

* Use of contact lenses in the last 3 months, or anticipated use of contact lenses during the study
* Cataract surgery, laser-assisted in situ keratomileusis [LASIK], or photorefractive keratectomy, within the last 6 months
* Current eye infection or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2015-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (10):
- United States (10):
  - North Bay Eye Associates, Petaluma, California
  - Eric M. White, OD, Inc., San Diego, California
  - Eye Center Northeast, Bangor, Maine
  - Moyes Eye Center, PC, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - David W. Ferris & Associates, Inc., Warwick, Rhode Island
  - Primary Eyecare Group, PC, Brentwood, Tennessee
  - The Eye Center at Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lievens C, Berdy G, Douglass D, Montaquila S, Lin H, Simmons P, Carlisle-Wilcox C, Vehige J, Haque S. Evaluation of an enhanced viscosity artificial tear for moderate to severe dry eye disease: A multicenter, double-masked, randomized 30-day study. Cont Lens Anterior Eye. 2019 Aug;42(4):443-449. doi: 10.1016/j.clae.2018.12.003. Epub 2018 Dec 17. PMID 30573298

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Started | 94 | 94
Completed | 93 | 91
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All 188 randomized patients were included in the Intent-to Treat (ITT) and safety populations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL® | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Customized [Number; unit: Participants]
  18 to less than 30 years | 11 | 13 | 24
  30 to 40 years | 11 | 14 | 25
  More than 40 years | 72 | 67 | 139
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Ocular Surface Disease Index© (OSDI©) Score
Description: The OSDI is a 12-question survey for patients to document their dry eye disease symptoms. The OSDI consists of a 5-point scale (0=none of the time and 4=all of the time), with higher scores representing greater disability. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability and 100=complete disability). A negative number change from baseline represents an improvement.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: All randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Number analyzed (Participants) | 94 | 94
Scores on a Scale
  Baseline | 42.44 (11.708) | 40.43 (11.232)
  Change from Baseline at Day 30 | -10.29 (15.864) | -7.48 (16.592)

2. Secondary Outcome: Change From Baseline in the OSDI© Score
Description: as for outcome 1
Time Frame: Baseline, Day 7
Population: Intent-to-Treat: All randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Number analyzed (Participants) | 94 | 94
Scores on a Scale
  Baseline | 42.44 (11.708) | 40.43 (11.232)
  Change from Baseline at Day 7 | -5.74 (14.338) | -2.34 (12.294)

3. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT)
Description: TBUT is the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement). The eye with shorter average TBUT at baseline is reported for each patient.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: All randomized patients
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Number analyzed (Participants) | 94 | 94
Seconds
  Baseline | 5.38 (1.674) | 5.40 (2.138)
  Change from Baseline at Day 30 (N-94, 93) | 0.84 (1.968) | 0.70 (4.139)

4. Secondary Outcome: Change From Baseline in the Combined Corneal and Conjunctival Staining Scores
Description: The cornea is the transparent front part of the eye which covers the iris and pupil. The conjunctiva is the clear membrane covering the white surface of the eye. The cornea is divided into 5 zones and the nasal and temporal conjunctiva is divided into 6 zones. The combined staining score is based on the sum of the five zones on the cornea and the six zones on the conjunctiva. Each zone is graded on a 0-5 scale (0=None; 1=trace; 2=mild; 3=moderate; 4=severe; 5=very severe), for a total score ranging from 0-55. The higher the score, the worse the dry eye condition. A negative number change from baseline represents a decrease in the severity of staining (improvement). The eye with higher score at baseline is reported for each subject.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: All randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Number analyzed (Participants) | 94 | 94
Scores on a Scale
  Baseline | 10.9 (7.24) | 11.8 (7.16)
  Change from Baseline at Day 30 (N=93, 91) | -1.7 (4.66) | -2.0 (6.12)

5. Secondary Outcome: Change From Baseline in the Schirmer Test
Description: The Schirmer's Test measures the rate of the secretion of tears produced by the eye over 5 minutes. The results indicate the presence of dry eye. The eye with the lower value at Baseline was used for Analysis. Normal = greater than or equal to 15 millimeters (mm) of tears, Dry Eye = less than 15 mm of tears.. The smaller the number, the more severe the dry eye. A positive number change from Baseline indicates improvement. The eye with the lower value at baseline is used for each subject.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: All randomized patients
Measure: Mean (Standard Deviation); unit: mm/5 min
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Number analyzed (Participants) | 94 | 94
mm/5 min
  Baseline | 9.98 (7.178) | 11.32 (8.496)
  Change from Baseline at Day 30 (N=88, 86) | 0.89 (5.601) | 0.69 (6.479)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from Screening through Day 30.
Description: The Safety Population included all patients who received at least 1 dose of the study treatment. The Safety Population was used to assess adverse events and serious adverse events.
Arm/Group | Refresh Optive® Gel Drops | REFRESH LIQUIGEL®
Serious Adverse Events (participants affected / at risk) | 0/94 | 1/94
Other Adverse Events (participants affected / at risk) | 7/94 | 5/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Refresh Optive® Gel Drops (N=94) | REFRESH LIQUIGEL® (N=94)
Hyphaema (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Refresh Optive® Gel Drops (N=94) | REFRESH LIQUIGEL® (N=94)
Vision blurred (Eye disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.